CLINICAL TRIAL: NCT02081235
Title: Incidence, Risk Factors, and Risk Model of Acute Kidney Injury in Pediatric Patients Who Undergoing Surgery for Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, WonHo Kim, Assistant Professor, Samsung Medical Center
Other Study IDs: 2013-12-101
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Patients Undergoing Surgery for Congenital Heart Disease
Keywords: congenital heart disease; acute kidney injury; risk factor; anesthesia
MeSH Terms: conditions — Heart Defects, Congenital; Acute Kidney Injury | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients who underwent surgery for congenital heart disease: patients who underwent surgery for congenital heart disease during 2012 in Samsung Medical Center
  Interventions: Procedure: surgery for congenital heart disease

INTERVENTIONS:
Procedure: surgery for congenital heart disease — surgery for congenital heart disease

SUMMARY:
Acute kidney injury (AKI) is a major complication after cardiac surgery and has been reported to be associated with adverse outcome. Previous studies have reported that the incidence of AKI in patients undergoing surgery for congenital heart disease is as high as 42% and AKI increase the patient mortality, intensive care unit stay and hospital stay. Previous studies have reported several risk factors for AKI after congenital heart surgery, however, perioperative variables including anesthesia-related factors have not been evaluated fully. Therefore, the investigators attempt to find out independent risk factors regarding perioperative variables.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a major complication after cardiac surgery and has been reported to be associated with adverse outcome. Previous studies have reported that the incidence of AKI in patients undergoing surgery for congenital heart disease is as high as 42% and AKI increase the patient mortality, intensive care unit stay and hospital stay. Previous studies have reported several risk factors for AKI after congenital heart surgery, however, perioperative variables including anesthesia-related factors have not been evaluated fully. In addition, a neutrophil-lymphocyte ratio (NLR), which have been reported to be a marker for systemic inflammation and associated with prognosis of cardiac and cancer patients might be able to predict development of postoperative AKI. Therefore, the investigators attempt to assess independent risk factors regarding perioperative variables including transfusion-related parameters, preoperative anemia, preoperative hypoalbuminemia, pulmonary hypertension, use of nitric oxide, use of hydroxyethyl starch, perioperative medication, hemodynamic variables and perioperative NLR.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent surgery for congenital heart disease between January 2012 and December 2012 in Samsung Medical Center

Exclusion Criteria:

* incomplete data for creatinine, estimated glomerular filtration rate, or urine output required to diagnose acute kidney injury
* patients who expired within 24 hours after surgery

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients who underwent surgery for congenital heart disease between 2009 and 2013 in Samsung Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury as defined by KDIGO (Kidney Disease: Improving Global outcome) criteria | during seven days after surgery
  Acute kidney injury as defined by KDIGO criteria (Stage 1, 2, 3)

SECONDARY OUTCOMES:
Acute kidney injury as defined by AKIN (acute kidney injury network) criteria | within 48 hours after surgery
  Acute kidney injury as defined by AKIN (acute kidney injury network) criteria within 48 hours after surgery
acute kidney injury diagnosis defined by RIFLE criteria | during seven days after surgery
  acute kidney injury diagnosis defined by RIFLE criteria (for Risk, Injury, Failure during seven days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea